CLINICAL TRIAL: NCT05819697
Title: FIRE Trial: Reducing Patient Memory Recall in the Burning Mouth Patient Population
Brief Title: Reducing Patient Memory Recall in the Burning Mouth Patient Population
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 843642
Record Dates: First submitted 2023-03-10; First posted 2023-04-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Burning Mouth Syndrome
Keywords: burning mouth syndrome; oral pain; burning mouth; chronic intraoral burning sensation
MeSH Terms: conditions — Burning Mouth Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FIRE Trial Participants: This study only has one group. All participants will receive the same intervention (smart phone app/texting notifications).
  Interventions: Other: FIRE Trial/Track Your Happiness notifications

INTERVENTIONS:
Other: FIRE Trial/Track Your Happiness notifications — All participants will receive notifications to their smart phones 3 times a day for 12 weeks. They will be asked questions related to burning mouth, to exercise as well as non-clinical Track Your Happiness questions, e.g., "Are you interacting with anyone right now?" "How do you feel right now?"

SUMMARY:
The goal of this study is to learn about burning mouth syndrome symptoms in real time in patients with burning mouth syndrome. The main questions it aims to answer are:

(1) To test the ability of a smartphone app to collect repeated observations of individual data to assess fluctuations in BMS symptoms (pain) at multiple points in the day as they happen; (2) To evaluate a panel of salivary biomarkers in patients with burning mouth syndrome (BMS) and to study their relationship with clinical variables. With a collaboration between Penn Dental Medicine and Wharton School of Business, our proposal aims to vastly improve the characterization of burning mouth syndrome through the use of a smartphone app and/or text-based notification.

Participants will attend 2 study visits where they will complete questionnaires and provide saliva samples and will respond to notifications/text message prompts on their smart phone 3 times a day for 12 weeks.

DETAILED DESCRIPTION:
This is a prospective study with the aims: (1) To test the ability of a smartphone app to collect repeated observations of individual data to assess fluctuations in BMS symptoms (pain) at multiple points in the day as they happen; (2) To evaluate a panel of salivary biomarkers in patients with burning mouth syndrome (BMS) and to study their relationship with clinical variables.

Participants will attend 2 study visits. Visit 1 of the study will consist of screening during the baseline visit. It will include administration of questionnaires, informed consent, collection of salivary samples, helping to download the app and/or helping to set up the smartphone to receive text notifications, and assisting with the demonstration of taking surveys on smartphones.

Track Your Happiness app, a smartphone and/or text-based notification system to take surveys, will collect data on people's experiences across a random sample of the moments of their lives. Participants will receives notifications 3 times per day at random times, and will be prompted to answer questions related to the burning mouth, to exercise, and a random selection of non-clinical Track Your Happiness questions, e.g., "Are you interacting with anyone right now?" "How do you feel right now?" Participants will receive these notifications for 12 weeks.

The final study visit (visit 2) will take place 12 weeks after Visit 1. Visit 2 will consist of questionnaires and collection of salivary samples.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 years and older
2. Willing and able to provide informed consent
3. Have been diagnosed with BMS for at least three months by an Oral Medicine or other specialist
4. Willing to submit a saliva sample
5. Have continuous access to a smartphone

Exclusion criteria:

1. In the opinion of the investigator, is unable or unlikely to comply fully with the study requirements or procedures for any reason (e.g. cognitive or physical impairment)
2. Prior head and neck radiation and/or chemotherapy
3. Medications that modulate or suppress the inflammatory system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will be patients who have been diagnosed with burning mouth syndrome by Oral Medicine specialists.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Track Your Happiness App utilization for Burning Mouth Syndrome (BMS) symptom reports in real time | 12 weeks
  Track Your Happiness app on smartphone and/or text base notification system will collect data in real time on people's experiences across a random sample of the moments of their lives through surveys. Participants will receive a notification on their phone at three random times each day and be prompted to answer questions adapted from the FIRE questionnaire related to burning mouth syndrome symptoms.

SECONDARY OUTCOMES:
Salivary Biomarkers | Baseline and follow up visit (12 weeks after baseline)
  The relationship between salivary biomarkers and burning mouth syndrome (BMS) symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Ko, DDS, Principal Investigator — Penn Dental School of Medicine, Center for Clinical and Translational Research
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT05819697/ICF_000.pdf